CLINICAL TRIAL: NCT01201512
Title: Primary Care Management for TMJD Pain
Brief Title: CONDOR Temporomandibular Muscle and Joint Disorders (TMJD) Survey
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other)
Responsible Party: Gregg H. Gilbert, DDS, MBA, Study Chair, The University of Alabama at Birmingham
Other Study IDs: 129134; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Temporomandibular Disorders
Keywords: TMJD pain; feasibility
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Temporomandibular disorders

SUMMARY:
The purpose of study was to characterize using an online questionnaire the feasibility of recruiting dentists in primary care dental practices in the practice-based research network and documenting their current initial care for their TMJD pain patients.

DETAILED DESCRIPTION:
The overall goal of this project was to collect data to be used in preparing an application for a Clinical Trial Planning Grant and then in designing a subsequent Phase III clinical trial. The ultimate goal of this series of research projects is to determine the most practical approach to conduct a randomized clinical trial (RCT) to evaluate initial intervention for patients with painful temporomandibular muscle and joint disorders (TMJD) using NIDCR's Collaboration of Networked Dental and Oral Health Research (CONDOR) group consisting of three dental Practice-Based Research Networks: The Dental Practice-Based Research Network (DPBNR), Northwest Practice-Based Research Collaborative in Evidence-based Dentistry (PRECEDENT), and Practitioners Engaged in Applied Research and Learning (PEARL).

ELIGIBILITY:
Inclusion Criteria:

* DPBRN dentist practitioner-investigator (general dentists or specialists) who had completed a DPBRN Enrollment Questionnaire
* 22 years of age or older

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The questionnaire was administered to all enrolled DPBRN dentist practitoner-investigators (general dentists or specialists), defined as those who had completed a DPBRN Enrollment Questionnaire who were 22 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg H Gilbert, DDS, MBA, Principal Investigator — The University of Alabama at Birmingham; Eric Schiffman, DDS, Study Chair — University of Minnesota
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- See also: Dental Practice-Based Research Network — http://DPBRN.org
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org